CLINICAL TRIAL: NCT06388265
Title: Emotional and Oral Characteristics of Patients That Attend a Dental Consultation for the Extraction of Third Molars
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Barcelona (Other)
Responsible Party: Principal Investigator, Mayra Schemel Suarez, Principal Investigator, University of Barcelona
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 18/2018, Acta 26-6-2018
Record Dates: First submitted 2024-04-20; First posted 2024-04-29 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Anxiety and Fear
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Verbal and Written detailed information (Experimental): The experimental group will receive verbal information about the procedure (exodontia of third molars) and additionally a trifold with detailed information about the surgical procedure.
  Interventions: Other: Trifold information
- Control (No Intervention): The control group will only receive verbal information about the surgical procedure.

INTERVENTIONS:
Other: Trifold information — Additional detailed and written information about the procedure will be given to the participants
  Arms: Verbal and Written detailed information

SUMMARY:
Analyze the level of anxiety, hemodynamic parameters, oral status, and satisfaction among patients undergoing third molar extraction, we will assess those who attend the Master of Oral Medicine, Surgery, and Implantology program at the University of Barcelona.

ELIGIBILITY:
Inclusion Criteria:

* Individuals 18 years old or older, from both genders that wished to voluntarily participate in the study and that required the extraction of third molars.

Exclusion Criteria:

* Systemic diseases (ASA III or IV) that contraindicate the performance of the surgical procedure
* Pregnant women
* Individuals that did not understand and/or could not respond the given questionnaire.
* Patients that required the extraction of a different tooth than a third molar or that required the extraction of more than two third molars in the same surgical time.
* Patients who had undergone extraction of a third molar in the twelve months prior to the current visit.
* Patients taking antidepressant medication or anxiolytic medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2022-01-09 (Actual); Primary Completion 2025-07-31 (Actual); Study Completion 2025-07-31 (Actual)

PRIMARY OUTCOMES:
Changes in STAI-S | Through study completion, an average of 5 weeks
  The Anxiety State scale (S-Anxiety) is an inventory that has been validated and assesses the current state of anxiety of the participant measured through an auto evaluation, asking how the evaluated individual feels "in this moment", using items that measure subjective feelings of apprehension, tension, nervousness, worry and activation/excitement of the autonomic nervous system.
  The total scores can go from 20 to 80 points A cut point value of 39 to 40 points has been suggested to detect clinically significant symptoms in the Anxiety State scale.
  STAI-S will be assessed in 4 stages:
  1. At the initial consultation (baseline)
  2. Immediately before the procedure and administration of the local anaesthetic solution
  3. Immediately after the procedure is completed
  4. 1 week after the procedure (exodontia)
Changes in MDAS | up to 3 weeks
  The modified dental anxiety scale (MDAS) is an auto evaluation questionnaire about dental anxiety that contains 5 items, each one with 5 possible answers that reflects in order an increase of anxiety (no anxiety to extremely anxious).
  The total score can go from 5 points to a maximum of 25 points. The lower limit to define an individual with extreme anxiety is 19 points and to define the presence of anxiety the score must be higher than 10 points.
  MDAS will be assessed in 2 stages:
  1. At the initial consultation (baseline)
  2. Immediately before the procedure and administration of the local anaesthetic solution

SECONDARY OUTCOMES:
Changes in blood pressure | Through study completion, an average of 5 weeks
  Changes in Blood pressure (Systolic and dyastolic) measured in mmHg
  Blood pressure will be assessed in 5 stages:
  1. At the initial consultation (baseline)
  2. Immediately before the procedure and administration of the local anaesthetic solution
  3. Immediately after administration of the local anaesthetic solution
  4. Immediately after the procedure is completed
Changes in Heart rate | Through study completion, an average of 5 weeks
  Changes in heart rate measured in beats per minute
  Heart rate will be assessed in 5 stages:
  1. At the initial consultation (baseline)
  2. Immediately before the procedure and administration of the local anaesthetic solution
  3. Immediately after administration of the local anaesthetic solution
  4. Immediately after the procedure is completed
Changes in Oxygen saturation | Through study completion, an average of 5 weeks
  Changes in oxygen saturation measured in percentage (%)
  Oxygen saturation will be assessed in 5 stages:
  1. At the initial consultation (baseline)
  2. Immediately before the procedure and administration of the local anaesthetic solution
  3. Immediately after administration of the local anaesthetic solution
  4. Immediately after the procedure is completed
Patient Satisfaction of procedure | 1 week after the procedure
  A questionnaire will be provided to the participants that consists of 6 questions, 2 questions to know the degree of discomfort at the last visit (suture removal control post exodontia) with 4 possible answers: none, little, moderate, a lot; and 4 questions to determine the degree of satisfaction with all the dental treatment carried out with affirmative or negative answers

CONTACTS AND LOCATIONS:
Overall Officials: José López-López, PhD, Study Director — University of Barcelona; Mayra Schemel Suarez, DDS, Principal Investigator — University of Barcelona
Locations (1):
- Hospital Odontològic Universitat de Barcelona, L'Hospitalet de Llobregat, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No